CLINICAL TRIAL: NCT02979652
Title: Can Point of Care Chest Ultrasound Predicts Pulmonary Complications After Major Surgery?
Acronym: POCUSR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Nord (Other)
Responsible Party: Sponsor
Other Study IDs: 00010254-2016 -016
Record Dates: First submitted 2016-11-24; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Intensive Care, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is done to estimate prevalence of the main detectable lung and cardiovascular complications by an ultrasound realized in room of post-interventional supervision at the patients whose duration of general anesthesia is superior at one hour after a surgery to risk

ELIGIBILITY:
Inclusion Criteria:

* Physical status score > 1
* Anesthesia of duration > 1 hour
* Visceral, orthopaedic, vascular, thoracic surgery, neurosurgery

Exclusion Criteria:

* Technical incapacity of accessibility to the ultrasound window
* Cardiac or pulmonary transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospatilized for a major surgery
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
cardiac and pulmonary functions | 1 hour
  cardiac and pulmonary functions will be evaluated by cardiac and pulmonary ultrasound exams for all patient whom have a more than 1 hour surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marc Leone, MD, Study Director — Departement anesthesie reanimation hopital nord
Locations (1):
- Departement anesthesie reanimation hopital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No